CLINICAL TRIAL: NCT01898533
Title: A Pilot Study of the Feasibility of Blood Oxygenation Level-Dependent Contrast ( BOLD) Breast MRI Induced by Breath- Holding
Brief Title: Feasibility of Blood Oxygenation Level-Dependent Contrast (BOLD) Breast MRI Induced by Breath- Holding
Acronym: BOLD
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00046072
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study, investigators intend to measure changes in BOLD contrast in the breast induced by breath-holding for subjects receiving radiation therapy to the breast. This study will provide the preliminary data and experience needed to successfully apply BOLD to quantify changes in oxygenation and blood flow of breast and tumor for a larger cohort of breast radiotherapy patients. The current study has the following objectives:

1. To determine the feasibility of BOLD contrast MRI of the breast, induced by breath-hold.
2. To measure the change in BOLD contrast of the breast and / or chest wall tissue for females undergoing radiotherapy

DETAILED DESCRIPTION:
11 subjects were consented to the trial. One subject voluntarily withdrew before any study procedures were performed.

ELIGIBILITY:
Inclusion Criteria: • Post-operative patients who are undergoing planning for future whole breast radiation therapy may be included in the study

* Female
* Age ≥18
* Negative serum pregnancy test for women of child bearing potential
* Signed study-specific informed consent

Exclusion Criteria:

* Unable to perform breath-holding of adequate duration.
* Unable to lie prone for approximately one hour during the study procedure
* Breast implants
* Any condition for which a MRI procedure is contraindicated including presence of metallic material in the body, such as pacemakers, non- MRI compatible surgical clips, shrapnel, etc.
* Positive serum pregnancy test
* Mastectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female subjects with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The change in BOLD contrast of the breasts and / or chest wall tissue will be measured by comparing breath hold sequences to normal breathing. | During MRI approx 1 hour
  Subjects will be evaluated holding their breath and during normal breathing.
Feasibility as measured by a BOLD contrast signal in at least 30% of subjects | During MRI approx one hour
  The imaging technique will be considered feasible if for any of the proposed imaging sequences, breath-holding induces a measurable (≥3× standard deviation of background) BOLD contrast signal in at least 30% of the subjects. Contrast will be measured by comparing breath hold sequences to normal breathing.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Blitzblau, MD PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States